CLINICAL TRIAL: NCT02926521
Title: Assessing Current Peripheral Nerve Block Catheter Fixation and Dressing Strategies: An Equivalence Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID 19 RELATED FACTORS
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Roland Brusseau, Instructor, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-P00021819
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Regional Anesthesia Morbidity
Keywords: nerve block catheter; catheter fixation; catheter dressing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dressing A (No Intervention): Dressing A: a nerve block catheter affixed with Pajunk anchor and covered with Tegaderm.
- Dressing B (Active Comparator): Dressing B: a nerve block catheter affixed with Pajunk anchor, skin treated with gum mastic liquid adhesive (Mastisol), all covered with Tegaderm
  Interventions: Device: Gum Mastic
- Dressing C (Active Comparator): Dressing C: a nerve block catheter sealed with 2-octyl cyanoacrylate liquid adhesive (Dermabond), trailing catheter affixed with Pajunk anchor, all covered with Tegaderm
  Interventions: Device: 2-octyl cyanoacrylate
- Dressing D (Active Comparator): Dressing D: a nerve block catheter sealed with 2-octyl cyanoacrylate (Dermabond), trailing catheter affixed with Pajunk anchor, skin treated with gum mastic liquid adhesive (Mastisol), all covered with Tegaderm
  Interventions: Device: 2-octyl cyanoacrylate; Device: Gum Mastic

INTERVENTIONS:
Device: 2-octyl cyanoacrylate — Addition of 2-octyl cyanoacrylate liquid adhesive to nerve catheter dressing
  Other Names: Dermabond
  Arms: Dressing C; Dressing D
Device: Gum Mastic — Addition of gum mastic liquid adhesive to nerve catheter dressing
  Other Names: Mastisol Liquid Adhesive
  Arms: Dressing B; Dressing D

SUMMARY:
The investigators' objective is to evaluate whether any of the various peripheral nerve block catheter dressing strategies currently employed by the Boston Children's Hospital Regional Anesthesia Service has any differential impact on specific outcome endpoints such as regional block catheter dislodgement, catheter occlusion, catheter leakage, skin irritation, and skin infection.

DETAILED DESCRIPTION:
Generally speaking, the goals of affixing and dressing a peripheral nerve block (PNB) catheter include preservation of the position and integrity of the catheter, the integrity of the skin, and avoidance of infection. In order to accomplish this, nerve block catheters at Boston Children's Hospital (BCH) are affixed to a patient's skin and dressed in a number of ways, usually based on provider preference.

Just as care providers routinely employ several combinations of tape, occlusive dressings and skin preparations to secure and protect intravenous catheters (all thought to be standard-of-care based on their frequency of use), so do the members of the regional service dress PNB catheters with various combinations of catheter anchors, Dermabond, Mastisol, and Tegaderms. The exact combinations are based on physician preference and/or habit, though all dressing schemes generally employ at minimum a standard catheter anchor (provided by the catheter manufacturer) and a Tegaderm, frequently with the addition of either Mastisol or Dermabond or both in combination. The four possible combinations in current use are:

1. Catheter anchor and Tegaderm only; 2. catheter anchor, Mastisol and Tegaderm; 3. catheter anchor, Dermabond and Tegaderm; 4. catheter anchor, Mastisol, Dermabond and Tegaderm

As no formal record is kept of dressing type and/or components, there is no accurate way of quantifying the frequencies of these dressing types being employed much less whether certain dressing strategies historically have been more effective than others maintaining the integrity of the catheter and surrounding skin.

These variations in routine practice suggest that there is not agreement about the benefits of adding either Mastisol or Dermabond (or both) to a dressing scheme, especially given their potential liabilities which include skin irritation (Mastisol, anecdotal at BCH), expense (Dermabond, approximately $20/use) and time (a couple of minutes drying time for each of these added elements).

Mastisol is a waterproof, clear liquid adhesive that has largely replaced tincture of benzoin as part of occlusive dressings (for nerve block catheters, IVs, arterial and central lines) as it is reported to have a significantly lower risk for skin irritation (1). As such, Mastisol has essentially become a standard of care for skin fixation and dressing of numerous catheter types. Papers in both the adult and pediatric regional anesthesia literature cite the use of Mastisol as a routine component of catheter fixation and dressing as well (2-4). However, there is little data in the literature evaluating the efficaciousness of Mastisol insofar as reducing catheter leakage or dislodgement and hence justifying its continued use as a part of catheter dressings. One study on healthy adults demonstrated differential forces required to dislodge a taped IV catheter with or without Mastisol (64 ± 1 vs. 46 ± 2 Newtons) however there is no data about catheter dislodgement rates over time in a clinical setting (5). One case report in the pediatric literature proposes a theoretical benefit of Mastisol use insofar as preventing regional anesthesia catheter dislodgement, but it too provides no clinical data (6).

Dermabond is a cyanoacrylate tissue adhesive that forms a strong bond across apposed wound edges, allowing normal healing to occur below and serving as a barrier to bacterial infiltration of the wound. It has been marketed to replace sutures that are 5-0 or smaller in diameter for incisional or laceration repair. This adhesive has been shown to save time during wound repair, to provide a flexible water-resistant protective coating and to eliminate the need for suture removal. Like Mastisol, Dermabond has become a commonplace addition to PNB catheter dressings for securement and puncture/insertion site closure both at BCH and nationally. And again, like Mastisol, there is little available data regarding whether Dermabond use as a part of the dressing scheme makes any difference insofar as catheter dislodgment or prevention of infection. A case series of three patients has been reported as recently as 2003 that described inclusion of Dermabond as a technique offering a simple, alternative method to secure a catheter for a prolonged period of time yet offered no qualitative or quantitative outcomes data (7). Other, more invasive, methods to fasten catheters have been advocated as well, such as suturing, retrograde subcutaneous tunneling (8), and cutaneous sutures (9).

Providers at BCH and elsewhere do not so much disagree as to what is the correct dressing for a nerve block catheter might be as they simply do not have relevant data to guide their decision-making. The physicians at BCH and at other institutions are using that method they believe is best by incorporating their own personal experiences as well as those of other clinicians. All agree that the primary goals, or benefits, of a good dressing system would be effective catheter stabilization, prevention of catheter occlusion or leakage, keeping the site clean and dry, and avoidance of infection. To-date, however, nerve block catheter dressings have not been studied in any rigorous way that might evaluate the various techniques for such outcomes.

There is scant literature available on this topic generally, despite a dressing's presumed importance in maintaining the appropriate position of the nerve block catheter and tip for maximal efficacy. The literature, if it can be called that, is largely comprised of numerous YouTube videos describing dressing and securing methodologies for nerve catheters (10); however none have been reported as having been evaluated in any rigorous prospective or retrospective analysis. (Reference to this general category of YouTube videos is made here as they essentially are a source of, and reflect, the standard of care and as such indicate the relative lack of rigorous evaluation of catheter securing techniques currently available).

Therefore the investigators wish to study whether the addition of Mastisol, Dermabond or both to PNB catheter dressings here at BCH has any influence on outcomes such as catheter dislodgment or function, skin integrity, and avoidance of infection. As such, the investigators propose a prospective, randomized study of equivalence of dressing type with the hypothesis that there is no more than a 10% difference in the rate of catheter dislodgement (the primary endpoint) between the 4 commonly used dressing schemes for PNB catheters at BCH.

ELIGIBILITY:
Inclusion Criteria:

* all subjects who are 0-100 years of age who are scheduled to receive a PNB catheter of one of the following types:

  * lumbar plexus
  * paravertebral
  * femoral
  * sciatic
  * brachial plexus (infraclavicular, supraclavicular and interscalene approach)
  * TAP (transversus abdominis plane)

Exclusion Criteria:

* Exclusions would be any patient with a known contraindication to any of the dressing materials and/or any block catheter that must be tunneled for clinical reasons.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
nerve block catheter dislodgement | duration of catheter use, up to but not longer than, 1 week
  presence or absence of catheter dislodgement (catheter out or no longer in a clinically effective position)

SECONDARY OUTCOMES:
nerve block catheter occlusion | duration of catheter use, up to but not longer than, 1 week
  presence or absence of catheter occlusion
nerve block catheter leakage | duration of catheter use, up to but not longer than, 1 week
  presence or absence of catheter leakage (presence of local anesthetic under occlusive dressing)
skin irritation at site of nerve block catheter skin entry | duration of catheter use, up to but not longer than, 1 week
  presence or absence of skin irritation (presence of hyperemic cutaneous reaction not present at dressing placement)
catheter site infection | duration of catheter use, up to but not longer than, 1 week
  presence or absence of catheter site infection (presence of purulent material)

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children"S Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No